CLINICAL TRIAL: NCT01969773
Title: Intravesical Botulinum Toxin A Injection in Treatment of Interstitial Cystitis Refractory to Conventional Treatment - A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Intravesical Botulinum Toxin A Injections in Treatment of Interstitial Cystitis Refractory to Conventional Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Director of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCGHUROL009
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Interstitial Cystitis
Keywords: Botulinum Toxin A (BoNT-A); Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: The patients were allocated to the treatment or control group by permuted block randomization code in a 2:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The attending doctors, patients, and study nurses did not know which solution was injected to their bladders, to keep the study in a double-blind condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum toxin A (Experimental): Patients will be randomly assigned to receive intravesical injection of 100U of BoNT-A (BOTOX, Allergan, Irvine, CA, USA)
  Interventions: Drug: Botulinum toxin A
- Control arm-Normal saline instillation (Placebo Comparator): Patients will be randomly assigned to receive intravesical injection of injection with normal saline.
  Interventions: Drug: Normal saline instillation

INTERVENTIONS:
Drug: Botulinum toxin A — Patients will be randomly assigned to receive intravesical injection of 100U of BoNT-A (BOTOX, Allergan, Irvine, CA, USA)
  Other Names: BoNT-A; BOTOX
  Arms: Botulinum toxin A
Drug: Normal saline instillation — Patients will be randomly assigned to receive intravesical injection of injection with normal saline.
  Other Names: N/S
  Arms: Control arm-Normal saline instillation

SUMMARY:
This study was designed in a multicenter, randomized, double-blind, placebo controlled trial to test the actual therapeutic effects of intravesical BoNTA injection. The results of this study might provide clinical evidence for a better therapeutic regimen in the treatment of IC/PBS.

DETAILED DESCRIPTION:
Background: Interstitial cystitis/painful bladder syndrome (IC/PBS) is a debilitating chronic disease of unknown etiology. Current treatments are usually unsuccessful in completely eradicating bladder pain and increasing bladder capacity. Although investigations on this topic have been enthusiastically performed, the etiology of IC/PBS remains unknown. Treatment based on single pathophysiology such as urothelial damage or neurogenic inflammation might not enough to eradicate the cascade of pathologies of IC/PBS.

Inhibition of neuroplasticity of the sensory fibers in the suburothelial space by intravesical BoNT-A injections might have good therapeutic targeting on pain and sensory urgency in patients with IC/PBS. In recent basic researches, BoNT-A has been shown to inhibit not only the release of acetylcholine and norepinephrine, but also that of nerve growth factor, adenosine triphosphate, substance P and calcitonin gene-related peptide from the nerve fibers and urothelium. This study was designed in a multicenter, randomized, double-blind, placebo controlled trial to test the actual therapeutic effects of intravesical BoNT-A injection on IC/PBS. The results of this study might provide clinical evidence for a better therapeutic regimen in the treatment of IC/PBS.

Materials and Methods: A total of 90 patients with IC/PBS who have failed conventional treatments for at least 6 months will be enrolled in this study. A diagnosis of IC/PBS has been established based on characteristic symptoms and cystoscopic findings of glomerulations, petechia, or mucosal fissures after hydrodistention. They will be investigated thoroughly on enrollment and will be excluded if not meeting the inclusion criteria of National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK). However, in this study the patients with Hunner's ulcer will not be included because previous study has shown that ulcer type IC/PBS does not respond to intravesical BoNT-A injection.

A 3-day voiding diary for functional bladder capacity, urinary frequency and nocturnal, O'Leary-Sant symptom and problem indexes, visual analog score (VAS), and videourodynamic parameters and potassium chloride (KCl) sensitivity test will be used to assess the therapeutic efficacy. Patients will be informed of the possible complications associated with BoNT-A injection such as generalized muscle weakness, difficult urination, transient urinary retention, or urinary tract infections. Eligible patients will be randomly assigned to receive intravesical injection of 100U of BoNT-A (BOTOX, Allergan, Irvine, CA, USA) (the treatment group) or injection with normal saline (control group). The intravesical injection will be performed immediately followed by cystoscopic hydrodistention under intravenous general anesthesia in the operation room.

Blood (10ml) and urine samples (30ml) will be collected before intravesical injection and after bladder hydrodistention. Bladder wall biopsies will also be performed after hydrodistention. The patients will be allocated to treatment or control group by the permuted block randomization code in 2:1 ratio, which is centrally controlled by a clinical pharmacist who prepares the solution for injection. Each vial of BoNT-A will be diluted with 10 ml of normal saline, resulting in 10U BoNT-A per 1.0 ml. Patients receive 20 suburothelial injections of BoNT-A solution or normal saline, each injection site receives 5U or saline in 0.5 ml. After the BoNT-A injections, patients will be followed up in the outpatient clinic 2 weeks and 4 weeks later. Then the patients will be followed up at out-patient clinic at 2 weeks, 4 weeks and 12 weeks. The primary end-point of this study is the reduction of bladder pain at 12-week follow-up. If patient has a reduction of VAS pain score of 2 or more, they will be considered as successfully treated. The treatment outcome will also be assessed by the global response assessment (GRA) to evaluate the overall perception of treatment result. The result will be considered as excellent when patients report improvement in the GRA by >2 or patients become free of bladder pain (VAS=0). Data will be compared between treatment and placebo groups. A p-value of less than 0.05 will be considered statistically significant.

Cystoscopy and bladder biopsy will be performed and sent for pathological examination and urological laboratory for investigations. The urine and serum biomarkers (NGF) and urothelial dysfunction markers (TUNEL for apoptosis, Ki-67 for proliferation, tryptase staining for mast cell activity, E-cadherin and zonula occludens-1 for junction protein expression) will be assessed to investigate the severity of urothelial dysfunction and chronic inflammation presented in these diseased bladders. Furthermore, the inflammatory protein assay such as TNFα, IL-6, IL-8 or TGF-beta will also be measured by protein array and western blotting. The urine and blood samples will be collected at baseline, 4 weeks, and end-point (12 weeks) in both treatment and controlled patients. The changes of urine and serum nerve growth factor (NGF) and cytokines (such as IL-1 beta, IL-6, IL-8, TNF-alpha) will be compared within group and between groups to provide laboratory evidence of decrease of bladder inflammation in IC/PBS. The changes of NGF and cytokines levels after BoNT-A injection treatments will also be compared in patients who respond and not respond to the treatment given. Urinary and serum NGF and cytokines levels were measured by the ELISA method.

Expected Results: The results of this study may demonstrate that intravesical injection of BoNT-A has a better clinical effect to provide greater pain relief and increase bladder capacity in patients with IC/PBS compared to the patients who received saline injection treatment. The clinical effect of BoNT-A on IC/PBS might be further reflected by the reduction of the serum or urinary NGF and cytokines levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IC/PBS who have failed conventional treatments for at least 6 months will be enrolled.
* A diagnosis of IC/PBS has been established based on characteristic symptoms and cystoscopic findings of glomerulations, petechia, or mucosal fissures after hydrodistention.
* All patients have been treated with at least two types of treatment modalities including non-steroid anti-inflammatory drugs, oral pentosan polysulfate sodium (PPS), intravesical instillation of heparin, hyaluronic acid, or tricyclic antidepressant for at least 6 months but the symptoms remained unchanged or relapsed.

Exclusion Criteria:

* Exclusion criteria proposed by NIDDK
* Automatic exclusions:

  1. Age <18 years old
  2. Benign or malignant bladder tumors
  3. Radiation cystitis Tuberculous cystitis
  4. Bacterial cystitis
  5. Vaginitis
  6. Cyclophosphamide cystitis
  7. Symptomatic urethral diverticulum
  8. Uterine, cervical, vaginal, or urethral cancer
  9. Active herpes
  10. Bladder or lower ureteral calculi
  11. Waking frequency <5 times in 12 hours
  12. Nocturia <2 times
  13. Symptoms relieved by antibiotics, urinary antiseptics, urinary analgesics (for example phenazopyridine hydrochloride)
  14. Duration < 12 months
  15. Involuntary bladder contractions (urodynamics)
  16. Capacity > 400ml, absence of sensory urgency
* Automatic inclusions:

  1.Hunner's ulcer
* Positive factors: (two positive factors are necessary for inclusion)

  1. Pain on bladder filling relieved by emptying
  2. Pain (suprapubic, pelvic, urethral, vaginal or peripheral)
  3. Glomerulations on endoscopy
  4. Decreased compliance on cystometrogram
  5. Bladder distention is defined arbitrarily as 80 cm water pressure for 1 minute
* Use of Anticholinergic drugs, for the treatment of lower urinary tract symptoms who have an effect.
* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up.
* Patients with bladder outlet obstruction on enrollment.
* Patients with urinary retention, PVR≥150 ml.
* Patients with uncontrolled confirmed diagnosis of acute urinary tract infection.
* Patients have laboratory abnormalities at screening including:

  1. Alanine aminotransferase (ALT) > 3 x upper limit of normal range
  2. Aspartate aminotransferase (AST) > 3 x upper limit of normal range.
  3. Patients have abnormal serum creatinine level > 2 x upper limit of normal range.
* Can not be used in the treatment of patients with transurethral catheter treatment.
* Pregnant and lactating women or women who intend to become pregnant during the study or have myasthenia gravis, Eaton Lambert syndrome.
* Patients with any other serious disease or condition considered by the investigator not suitable for entry into the trial.
* Patients participated investigational drug trial within 1 month before entering this study.
* Written informed consent has been obtained.
* Patient who did not complete the 3-day micturition diary according to the instruction.
* Intestinal bladder augmentation patients receive angioplasty for the treatment of overactive bladder.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Net change of Patient Perception of Visual Analogue Scale (VAS) | Baseline and 8 weeks
  Efficacy:
  The primary end-point of this study is the reduction of bladder pain at 8-week follow-up. If patient has a reduction of VAS pain score of 2 or more, they will be considered as successfully treated at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events

SECONDARY OUTCOMES:
Net change of Patient Perception of global response assessment (GRA) | Baseline and 8 weeks
  Efficacy:
  The treatment outcome will be assessed by the global response assessment (GRA) to evaluate the overall perception of treatment resultant at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of O'Leary-Sant symptom and problem indexes | Baseline and 8 weeks
  Efficacy:
  The IC symptoms will be assessed by the O'Leary-Sant symptom and problem indexes at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the functional bladder capacity (FBC) | Baseline and 8 weeks
  Efficacy:
  Patients will be requested to keep a 3-day voiding diary prior to treatment to record the functional bladder capacity (FBC). Then the patients will be followed up at out-patient clinic at 8 weeks.
  Safety:
  Systemic adverse events
Net change of the number of urinary frequency | Baseline and 8 weeks
  Efficacy:
  Patients will be requested to keep a 3-day voiding diary prior to treatment to record the number of urinary frequency at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the number of nocturnal | Baseline and 8 weeks
  Efficacy:
  Patients will be requested to keep a 3-day voiding diary prior to treatment to record the number of nocturnal at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the Quality of Life (QoL) | Baseline and 8 weeks
  Efficacy:
  Efficacy measured the net change of the Quality of Life (QoL) at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the maximal flow rate (Qmax) | Baseline and 8 weeks
  Efficacy:
  Efficacy measured the net change of the maximal flow rate (Qmax) at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the voided volume | Baseline and 8 weeks
  Efficacy:
  Efficacy measured the net change of the voided volume at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the residual urine volume (PVR) | Baseline and 8 weeks
  Efficacy:
  Efficacy measured the net change of the residual urine volume (PVR) at baseline and 8 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD was not planned to share

REFERENCES:
- [Background] Hanno PM, Sant GR. Clinical highlights of the National Institute of Diabetes and Digestive and Kidney Diseases/Interstitial Cystitis Association scientific conference on interstitial cystitis. Urology. 2001 Jun;57(6 Suppl 1):2-6. doi: 10.1016/s0090-4295(01)01112-8. PMID 11378041
- [Background] Payne CK, Mosbaugh PG, Forrest JB, Evans RJ, Whitmore KE, Antoci JP, Perez-Marrero R, Jacoby K, Diokno AC, O'Reilly KJ, Griebling TL, Vasavada SP, Yu AS, Frumkin LR; ICOS RTX Study Group (Resiniferatoxin Treatment for Interstitial Cystitis). Intravesical resiniferatoxin for the treatment of interstitial cystitis: a randomized, double-blind, placebo controlled trial. J Urol. 2005 May;173(5):1590-4. doi: 10.1097/01.ju.0000154631.92150.ef. PMID 15821499
- [Background] Nickel JC, Barkin J, Forrest J, Mosbaugh PG, Hernandez-Graulau J, Kaufman D, Lloyd K, Evans RJ, Parsons CL, Atkinson LE; Elmiron Study Group. Randomized, double-blind, dose-ranging study of pentosan polysulfate sodium for interstitial cystitis. Urology. 2005 Apr;65(4):654-8. doi: 10.1016/j.urology.2004.10.071. PMID 15833501
- [Background] Sant GR, Propert KJ, Hanno PM, Burks D, Culkin D, Diokno AC, Hardy C, Landis JR, Mayer R, Madigan R, Messing EM, Peters K, Theoharides TC, Warren J, Wein AJ, Steers W, Kusek JW, Nyberg LM; Interstitial Cystitis Clinical Trials Group. A pilot clinical trial of oral pentosan polysulfate and oral hydroxyzine in patients with interstitial cystitis. J Urol. 2003 Sep;170(3):810-5. doi: 10.1097/01.ju.0000083020.06212.3d. PMID 12913705
- [Background] Hanno PM, Buehler J, Wein AJ. Use of amitriptyline in the treatment of interstitial cystitis. J Urol. 1989 Apr;141(4):846-8. doi: 10.1016/s0022-5347(17)41029-9. PMID 2926877
- [Background] Sairanen J, Forsell T, Ruutu M. Long-term outcome of patients with interstitial cystitis treated with low dose cyclosporine A. J Urol. 2004 Jun;171(6 Pt 1):2138-41. doi: 10.1097/01.ju.0000125139.91203.7a. PMID 15126772
- [Background] Brady CM, Apostolidis AN, Harper M, Yiangou Y, Beckett A, Jacques TS, Freeman A, Scaravilli F, Fowler CJ, Anand P. Parallel changes in bladder suburothelial vanilloid receptor TRPV1 and pan-neuronal marker PGP9.5 immunoreactivity in patients with neurogenic detrusor overactivity after intravesical resiniferatoxin treatment. BJU Int. 2004 Apr;93(6):770-6. doi: 10.1111/j.1464-410X.2003.04722.x. PMID 15049988
- [Background] Cockayne DA, Hamilton SG, Zhu QM, Dunn PM, Zhong Y, Novakovic S, Malmberg AB, Cain G, Berson A, Kassotakis L, Hedley L, Lachnit WG, Burnstock G, McMahon SB, Ford AP. Urinary bladder hyporeflexia and reduced pain-related behaviour in P2X3-deficient mice. Nature. 2000 Oct 26;407(6807):1011-5. doi: 10.1038/35039519. PMID 11069181
- [Background] Beltinger J, McKaig BC, Makh S, Stack WA, Hawkey CJ, Mahida YR. Human colonic subepithelial myofibroblasts modulate transepithelial resistance and secretory response. Am J Physiol. 1999 Aug;277(2):C271-9. doi: 10.1152/ajpcell.1999.277.2.C271. PMID 10444403
- [Background] Cayan S, Coskun B, Bozlu M, Acar D, Akbay E, Ulusoy E. Botulinum toxin type A may improve bladder function in a rat chemical cystitis model. Urol Res. 2003 Feb;30(6):399-404. doi: 10.1007/s00240-002-0291-0. Epub 2003 Jan 21. PMID 12599022
- [Background] Steers WD, Tuttle JB. Mechanisms of Disease: the role of nerve growth factor in the pathophysiology of bladder disorders. Nat Clin Pract Urol. 2006 Feb;3(2):101-10. doi: 10.1038/ncpuro0408. PMID 16470209
- [Background] Apostolidis A, Popat R, Yiangou Y, Cockayne D, Ford AP, Davis JB, Dasgupta P, Fowler CJ, Anand P. Decreased sensory receptors P2X3 and TRPV1 in suburothelial nerve fibers following intradetrusor injections of botulinum toxin for human detrusor overactivity. J Urol. 2005 Sep;174(3):977-82; discussion 982-3. doi: 10.1097/01.ju.0000169481.42259.54. PMID 16094018
- [Background] Reitz A, Stohrer M, Kramer G, Del Popolo G, Chartier-Kastler E, Pannek J, Burgdorfer H, Gocking K, Madersbacher H, Schumacher S, Richter R, von Tobel J, Schurch B. European experience of 200 cases treated with botulinum-A toxin injections into the detrusor muscle for urinary incontinence due to neurogenic detrusor overactivity. Eur Urol. 2004 Apr;45(4):510-5. doi: 10.1016/j.eururo.2003.12.004. PMID 15041117
- [Background] Smith CP, Radziszewski P, Borkowski A, Somogyi GT, Boone TB, Chancellor MB. Botulinum toxin a has antinociceptive effects in treating interstitial cystitis. Urology. 2004 Nov;64(5):871-5; discussion 875. doi: 10.1016/j.urology.2004.06.073. PMID 15533466
- [Background] Kuo HC. Preliminary results of suburothelial injection of botulinum a toxin in the treatment of chronic interstitial cystitis. Urol Int. 2005;75(2):170-4. doi: 10.1159/000087173. PMID 16123573
- [Background] Giannantoni A, Costantini E, Di Stasi SM, Tascini MC, Bini V, Porena M. Botulinum A toxin intravesical injections in the treatment of painful bladder syndrome: a pilot study. Eur Urol. 2006 Apr;49(4):704-9. doi: 10.1016/j.eururo.2005.12.002. Epub 2006 Jan 4. PMID 16417964
- [Background] Rapp DE, Turk KW, Bales GT, Cook SP. Botulinum toxin type a inhibits calcitonin gene-related peptide release from isolated rat bladder. J Urol. 2006 Mar;175(3 Pt 1):1138-42. doi: 10.1016/S0022-5347(05)00322-8. PMID 16469640
- [Background] Chuang YC, Yoshimura N, Huang CC, Chiang PH, Chancellor MB. Intravesical botulinum toxin a administration produces analgesia against acetic acid induced bladder pain responses in rats. J Urol. 2004 Oct;172(4 Pt 1):1529-32. doi: 10.1097/01.ju.0000137844.77524.97. PMID 15371885
- [Background] Giannantoni A, Di Stasi SM, Nardicchi V, Zucchi A, Macchioni L, Bini V, Goracci G, Porena M. Botulinum-A toxin injections into the detrusor muscle decrease nerve growth factor bladder tissue levels in patients with neurogenic detrusor overactivity. J Urol. 2006 Jun;175(6):2341-4. doi: 10.1016/S0022-5347(06)00258-8. PMID 16697870
- [Background] Khera M, Somogyi GT, Kiss S, Boone TB, Smith CP. Botulinum toxin A inhibits ATP release from bladder urothelium after chronic spinal cord injury. Neurochem Int. 2004 Dec;45(7):987-93. doi: 10.1016/j.neuint.2004.06.001. PMID 15337297
- [Background] Kuo HC. Clinical effects of suburothelial injection of botulinum A toxin on patients with nonneurogenic detrusor overactivity refractory to anticholinergics. Urology. 2005 Jul;66(1):94-8. doi: 10.1016/j.urology.2005.02.002. PMID 15992869
- [Background] Cui M, Khanijou S, Rubino J, Aoki KR. Subcutaneous administration of botulinum toxin A reduces formalin-induced pain. Pain. 2004 Jan;107(1-2):125-33. doi: 10.1016/j.pain.2003.10.008. PMID 14715398
- [Background] Giannantoni A, Porena M, Costantini E, Zucchi A, Mearini L, Mearini E. Botulinum A toxin intravesical injection in patients with painful bladder syndrome: 1-year followup. J Urol. 2008 Mar;179(3):1031-4. doi: 10.1016/j.juro.2007.10.032. Epub 2008 Jan 18. PMID 18206941
- [Background] Lubeck DP, Whitmore K, Sant GR, Alvarez-Horine S, Lai C. Psychometric validation of the O'leary-Sant interstitial cystitis symptom index in a clinical trial of pentosan polysulfate sodium. Urology. 2001 Jun;57(6 Suppl 1):62-6. doi: 10.1016/s0090-4295(01)01126-8. PMID 11378052
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Vizzard MA. Changes in urinary bladder neurotrophic factor mRNA and NGF protein following urinary bladder dysfunction. Exp Neurol. 2000 Jan;161(1):273-84. doi: 10.1006/exnr.1999.7254. PMID 10683293
- [Background] Parsons CL, Housley T, Schmidt JD, Lebow D. Treatment of interstitial cystitis with intravesical heparin. Br J Urol. 1994 May;73(5):504-7. doi: 10.1111/j.1464-410x.1994.tb07634.x. PMID 8012771
- [Background] Chung SD, Kuo YC, Kuo HC. Intravesical onabotulinumtoxinA injections for refractory painful bladder syndrome. Pain Physician. 2012 May-Jun;15(3):197-202. PMID 22622903
- [Background] Seki S, Erickson KA, Seki M, Nishizawa O, Igawa Y, Ogawa T, de Groat WC, Chancellor MB, Yoshimura N. Elimination of rat spinal neurons expressing neurokinin 1 receptors reduces bladder overactivity and spinal c-fos expression induced by bladder irritation. Am J Physiol Renal Physiol. 2005 Mar;288(3):F466-73. doi: 10.1152/ajprenal.00274.2004. PMID 15692058
- [Background] Dell JR, Parsons CL. Multimodal therapy for interstitial cystitis. J Reprod Med. 2004 Mar;49(3 Suppl):243-52. PMID 15088863
- [Background] Liu HT, Kuo HC. Intravesical botulinum toxin A injections plus hydrodistension can reduce nerve growth factor production and control bladder pain in interstitial cystitis. Urology. 2007 Sep;70(3):463-8. doi: 10.1016/j.urology.2007.04.038. PMID 17905097
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597